CLINICAL TRIAL: NCT02288936
Title: Phase II Multicenter Study to Analyze the Predictive Value of Fusion Gene TMPRSS2-ETS in Response to Enzalutamide in Patients With Metastatic CRPC no Previously Treated With Chemotherapy
Brief Title: Analyze the Predictive Value of Gene TMPRSS2-ETS in Response to Enzalutamide in Patients With Prostate Cancer
Acronym: PREMIERE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Astellas Pharma Inc (Industry); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOG-MIE-2014-04; 2014-003192-28 (EudraCT Number)
Record Dates: First submitted 2014-10-28; First posted 2014-11-13 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Hormone-refractory Prostate Cancer
Keywords: Hormone-refractory prostate cancer; Enzalutamide; TMPRSS2-ETS fusion gene
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzalutamide (Experimental): Enzalutamide 160 mg/day
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide 160 mg/day

SUMMARY:
Prostate cancer is the most common non-skin tumor diagnosed in men and the second leading cause of cancer death in men in Western countries.

Between 10-20% of patients are diagnosed at metastatic stage and about half of those diagnosed in early stages will develop metastases.

After the clinical benefit of mitoxantrone and the improved survival of 2-3 months provided by docetaxel in first line, the second search is driven to look for effective second lines treatments. In recent years, there are new drugs for the treatment of prostate cancer, revolutionizing the therapeutic sequence and survival.

Thus, androgen deprivation therapy, treatment of choice, induces an improvement of symptoms in approximately 70-80% of patients, but it is limited by the development of mechanisms of resistance to androgen deficiency. Docetaxel was the first chemotherapy drug to increase survival in patients with metastatic prostate cancer. The second cytotoxic drug approved in the second line treatment of metastatic CRPC has been cabazitaxel.

Enzalutamide improves survival in patients with metastatic CRPC who had progressed to chemotherapy and also in patients who had not received chemotherapy.

To date, there are no biomarkers available that allow us to identify which patients from a clinical or molecular view are those that will be able to benefit from the treatment options currently available. The presence of the TMPRSS2-ETS rearrangement has been shown to correlate with efficacy in clinical practice abiraterone.

There is scientific and preclinical background that makes one suspect that the molecular alteration may influence the same way enzalutamide antiandrogen activity, but it has not been determined to date.

The objective of this study is to determine whether the efficacy and safety of enzalutamide, when administered to patients with castration resistant prostate cancer prior to administration of docetaxel is influenced by the presence or absence of the fusion gene TMPRSS2- ETS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above, willing and able to provide written informed consent.
* Prostate adenocarcinoma with histological or cytological confirmation without neuroendocrine differentiation nor small cell characteristics
* Androgen deprivation therapy with GnRH analogs or bilateral orchiectomy (pharmacological or surgical castration). Patients without bilateral orchiectomy must follow a GnRH analog therapy during the trial.
* Testosterone serum level <= 1,73 nmol/L (50 ng/dL) in screening visit.
* Patients under bisphosphonate therapy must have received stable doses for the last 4 weeks.
* Progression disease at inclusion, defined by one or more of the following three criteria during androgen deprivation therapy (according with the criterion nº 3): - PSA progression defined as two elevation of the PSA serum level with >=1 week between each measure. Patients who have received an antiandrogen must present disease progression (>=4 weeks since the last dose of flutamide or >=6 weeks since the last dose of bicalutamide or nilutamide). PSA value in screening visit must be >=2 μg/L (2 ng/mL). - Soft tissue progression defined by RECIST 1.1 criteria - Bone lesion progression defined by PCWG2 criteria, with two or more new lesions in a scintigraphy
* Metastatic disease with bone lesions detected by scintigraphy, or measurable soft tissue lesions by CT/MR. Patients with ganglionar disease will be suitable if they have at least one ganglionar lesion with smallest diameter > 2,5 cm.
* Patients without previous cytotoxic chemotherapy for prostate cancer
* Patients without previous abiraterone acetate therapy for prostate cancer - - Asymptomatic patient or mild symptomatic about prostate cancer, (answer in the question nº 3 of the Brief Pain Inventory Short From < 4) 11. ECOG = 0-1.
* Life expectancy of at least 6 months
* Patient must be able to swallow the investigation product and to follow the protocol requirements.
* Biomarker study informed consent

Exclusion Criteria:

* Active infection or other medical condition which, in the opinion of the investigator, would preclude participation in this trial.
* Known brain metastasis or leptomeningeal active involvement
* Other malignancy in the last five years, except non-melanoma skin cancer treated and resolved.
* Hematologic parameters: - Absolute neutrophil count <=1500/μL - Platelet count <100 000/μL - Haemoglobin < 5,6 mmol/L (9 g/dL)
* Liver function: Serum bilirubin, SGPT/ALT or SGOT/AST > 2,5 x ULN
* Renal function: Creatinine >177 μmol/L (2 mg/dL).
* Serum albumin <30 g/L (3,0 g/dL)
* History of epilepsy or other medical condition which could cause an epileptic crisis as syncope or transient ischemic attack in the last twelve months.
* Clinically significant cardiovascular disease.
* Known gastrointestinal (GI) disease that could interfere with the GI absorption.
* Significant surgery within 4 weeks before enrollment.
* Use of opioids to control cancer pain within 4 weeks before enrollment.
* Radiation therapy for treatment of the primary tumor in the last 3 weeks before enrollment
* Radiation therapy for treatment of metastases in the last two months
* Radionuclide therapy for treatment of bone metastasis
* Prior flutamide treatment within 4 weeks before enrollment
* Bicalutamide or nilutamide therapy within 6 weeks before enrollment
* 5-a reductase inhibitors, estrogen o cyproterone therapy within 4 weeks before enrollment
* Biologic therapy or other antitumoral drugs for the treatment of CRPC in the last 4 weeks
* History of cancer progression with ketoconazole
* Prior therapy or enrollment in a trial with an investigational product which blocks androgen synthesis (abiraterone, TAK-700, TAK-683, TAK-448) or blocks androgen receptors (ARN507, BMS 641988).
* Included in a previous trial with enzalutamide (MDV3100).
* Administration of an investigational drug in the last 4 weeks before enrollment
* Use of phytotherapy products which hormonal activity against prostate cancer or which reduce PSA levels, or systemic corticosteroids in a dose greater than the equivalent of prednisone 10mg/day, within 4 weeks before enrollment
* Hereditary fructose intolerance
* Any condition which, in the opinion of the investigator, would preclude participation in this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
PSA progression free survival | Up to 18 months
  Evaluate PSA progression (PCWG2 criteria) from date of patient inclusion until the date of first documented PSA progression or date of death from any cause, whichever came first, assessed up to 18 months.

SECONDARY OUTCOMES:
Number of individual events (hematologic events and not hematologic events) per patient | Up to 12 months
  Number of events per patient
Time to PSA response | Up to 18 months
  Time from start of treatment to PSA progression (PCWG2 criteria)
PSA response rate | Up to 18 months
  PSA response according to PCWG2 criteria, as % of patients with PSA response
Radiologic progression free survival | Up to 18 months
  Radiologic progression free survival according RECIST 1.1 criteria, from date of patient inclusion until the date of first documented radiologic progression or date of death from any cause, whichever came first, assessed up to 18 months.
Soft tissue response | Up to 18 months
  Soft tissue response according RECIST 1.1 criteria
Time until the beginning of cytotoxic chemotherapy | Up to 18 months
  Time from date of patient inclusion until the date of the start of cytotoxic chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Grande, MD, Study Director — Hospital Universitario Ramon y Cajal
Locations (16):
- Spain (16):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias I Pujol de Badalona, Badalona, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Parc Taulí, Barcelona
  - Complejo Hospitalario Regional Reina Sofía, Córdoba
  - Complejo Asistencial Universitario de Leon, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Hospitalario de Especialidades Virgen de La Victoria, Málaga
  - Hospital General Universitario J.M. Morales Meseguer, Murcia
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Complejo Hospitalario Regional Virgen Del Rocio, Seville
  - Fundación Instituto Valenciano de Oncologia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Jayaram A, Wingate A, Wetterskog D, Conteduca V, Khalaf D, Sharabiani MTA, Calabro F, Barwell L, Feyerabend S, Grande E, Martinez-Carrasco A, Font A, Berruti A, Sternberg CN, Jones R, Lefresne F, Lahaye M, Thomas S, Joshi S, Shen D, Ricci D, Gormley M, Merseburger AS, Tombal B, Annala M, Chi KN, De Giorgi U, Gonzalez-Billalabeitia E, Wyatt AW, Attard G. Plasma Androgen Receptor Copy Number Status at Emergence of Metastatic Castration-Resistant Prostate Cancer: A Pooled Multicohort Analysis. JCO Precis Oncol. 2019 Sep 24;3:PO.19.00123. doi: 10.1200/PO.19.00123. eCollection 2019. PMID 32923850
- [Derived] Wu A, Cremaschi P, Wetterskog D, Conteduca V, Franceschini GM, Kleftogiannis D, Jayaram A, Sandhu S, Wong SQ, Benelli M, Salvi S, Gurioli G, Feber A, Pereira MB, Wingate AM, Gonzalez-Billalebeitia E, De Giorgi U, Demichelis F, Lise S, Attard G. Genome-wide plasma DNA methylation features of metastatic prostate cancer. J Clin Invest. 2020 Apr 1;130(4):1991-2000. doi: 10.1172/JCI130887. PMID 32149736
- [Derived] Conteduca V, Wetterskog D, Sharabiani MTA, Grande E, Fernandez-Perez MP, Jayaram A, Salvi S, Castellano D, Romanel A, Lolli C, Casadio V, Gurioli G, Amadori D, Font A, Vazquez-Estevez S, Gonzalez Del Alba A, Mellado B, Fernandez-Calvo O, Mendez-Vidal MJ, Climent MA, Duran I, Gallardo E, Rodriguez A, Santander C, Saez MI, Puente J, Gasi Tandefelt D, Wingate A, Dearnaley D; PREMIERE Collaborators; Spanish Oncology Genitourinary Group; Demichelis F, De Giorgi U, Gonzalez-Billalabeitia E, Attard G. Androgen receptor gene status in plasma DNA associates with worse outcome on enzalutamide or abiraterone for castration-resistant prostate cancer: a multi-institution correlative biomarker study. Ann Oncol. 2017 Jul 1;28(7):1508-1516. doi: 10.1093/annonc/mdx155. PMID 28472366